CLINICAL TRIAL: NCT04991896
Title: Acute Management of Paroxysmal Atrial Fibrillation With Beta Blockers Plus Intravenous Flecainide: a Real-world Chios Registry (BETAFLEC-CHIOS)
Brief Title: Beta Blockers Plus Intravenous Flecainide for Paroxysmal Atrial Fibrillation: a Real-world Chios Registry (BETAFLEC-CHIOS)
Acronym: BETAFLEC-CHIOS
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Collaborators: Skylitseio General Hospital (Unknown)
Responsible Party: Principal Investigator, Matthaios Didagelos, Principal Investigator, Consultant Cardiologist, AHEPA University Hospital
Other Study IDs: 80-28/07/2021
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Sotalol; Bisoprolol; Metoprolol; Betaxolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Flecainide Injectable Product — Flecainide is given as an IV infusion of 1.5 mg/kg (max 150 mg) in DW 5% over 10 min under continuous monitoring. Concomitant administration of a b-blocker is also applied in all patients. The dose and type of b-blocker are selected according to heart rate during the AF and patient's medical history.
  Other Names: Sotalol, Bisoprolol, Metoprolol, Betaxolol

SUMMARY:
BETAFLEC-CHIOS, is a single-center registry that was initiated in the "Skylitseion" General Hospital of Chios in January 2020 and is ongoing. The inclusion criterion is IV flecainide administration for recent-onset AF lasting less than 48 hours. Oral b-blockers are co-administered in all patients. The main exclusion criteria are severe structural or ischemic heart disease and conduction system dysfunction. Continuous monitoring is applied during and after administration of IV flecainide. If no conversion to sinus rhythm is achieved at 2 hours after flecainide infusion, the patient is recorded as "unsuccessful conversion attempt".

DETAILED DESCRIPTION:
Patient population BETAFLEC-CHIOS, is a single-center registry that was initiated in the "Skylitseion" General Hospital of Chios in January 2020 and is ongoing. Patients are included in the registry if presenting with recent-onset atrial fibrillation (AF) (≤48 hours of onset) and lasting ≥30min, documented by a 12-lead ECG and having received intravenous (IV) flecainide on treating physician's discretion. Exclusion criteria are severe structural or ischemic heart disease (previous cardiac surgery, any cardiomyopathy, myocardial infarction at any time), atrial flutter, sick sinus syndrome, high degree atrioventricular block, bifascicular block, abnormal electrolyte levels (especially hypo- or hyperkalemia) or known sensitivity to flecainide. Continuous monitoring is applied during and after administration of IV flecainide. If no conversion to sinus rhythm is achieved at 2 hours after flecainide infusion initiation, the patient is recorded as "unsuccessful conversion attempt" and forwarded for direct current cardioversion (DCC). All patients were anticoagulated according to the current European Society Guidelines (ESC) or the management of AF [ESC Afib 2020].

Flecainide administration Flecainide is given as an IV infusion of 1.5 mg/kg (max 150 mg) in DW 5% over 10 min under continuous monitoring. Concomitant administration of a b-blocker is also applied in all patients. The dose and type of b-blocker are selected according to heart rate during the AF and patient's medical history. "Time to conversion" is calculated as the time interval from the end of the infusion up to when sinus rhythm is observed on the monitor and confirmed subsequently with a 12-lead ECG.

ELIGIBILITY:
Inclusion Criteria:

1. Informed written consent.
2. Recent-onset atrial fibrillation (AF) (≤48 hours of onset) and lasting ≥30min, documented by a 12-lead ECG
3. Administration of intravenous flecainide
4. Administration of an oral b-blocker

Exclusion Criteria:

1. Age <18 years
2. Severe structural or ischemic heart disease (previous cardiac surgery, any cardiomyopathy, myocardial infarction at any time)
3. Atrial flutter, sick sinus syndrome, high degree atrioventricular block, bifascicular block
4. Abnormal electrolyte levels (especially hypo- or hyperkalemia)
5. Known sensitivity to flecainide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are included in the registry if presenting with recent-onset atrial fibrillation (AF) (≤48 hours of onset) and lasting ≥30min, documented by a 12-lead ECG and having received intravenous (IV) flecainide on treating physician's discretion. Exclusion criteria are severe structural or ischemic heart disease (previous cardiac surgery, any cardiomyopathy, myocardial infarction at any time), atrial flutter, sick sinus syndrome, high degree atrioventricular block, bifascicular block, abnormal electrolyte levels (especially hypo- or hyperkalemia) or known sensitivity to flecainide. Continuous monitoring is applied during and after administration of IV flecainide.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients converted to sinus rhythm at 1 hour | 1 hour
  Successful cardioversion from atrial fibrillation to sinus rhythm at 1 hour

SECONDARY OUTCOMES:
Number of patients converted to sinus rhythm at 2 hour | 2 hours
  Successful cardioversion from atrial fibrillation to sinus rhythm at 2 hours
Number of patients with any documented proarrhythmic event | 2 hours
  Ventricular tachycardia, ventricular fibrillation, torsades de pointes, atrial flutter with 1:1 atrioventricular conduction
Number of arrhythmic events managed with defibrillation | 2 hours
  Any arrhythmic event managed with defibrillation
Number of patients with documented severe hypotension | 2 hours
  Systolic blood pressure <90 mmHg for >10 min or requiring inotropic support
Number of patients that discontinued IV flecainide infusion | 2 hours
  Discontinuation of the IV flecainide infusion for any reason
Hospitalization duration | 48 hours
  Total length of hospitalization duration in hours

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Kartalis, Principal Investigator — Skylitseio General Hospital of Chios; Matthaios Didagelos, Principal Investigator — AHEPA University General Hospital
Locations (1):
- Skylitseio General Hospital, Chios, Greece

IPD SHARING:
Plan to Share IPD: No